CLINICAL TRIAL: NCT01864746
Title: Phase III Study Evaluating Palbociclib (PD-0332991), a Cyclin-Dependent Kinase (CDK) 4/6 Inhibitor in Patients With Hormone-receptor-positive, HER2-normal Primary Breast Cancer With High Relapse Risk After Neoadjuvant Chemotherapy "PENELOPEB"
Brief Title: A Study of Palbociclib in Addition to Standard Endocrine Treatment in Hormone Receptor Positive Her2 Normal Patients With Residual Disease After Neoadjuvant Chemotherapy and Surgery
Acronym: PENELOPE-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Pfizer (Industry); AGO Study Group (Other); NSABP Foundation Inc (Network); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBG78/BIG 1-13/NSABP-B-54-I; 2013-001040-62 (EudraCT Number)
Record Dates: First submitted 2013-05-14; First posted 2013-05-30 (Estimated); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Hormonreceptor Positive; Her2-normal; Postneoadjuvant Treatment With CDK 4/6 Inhibitor; CPS-EG Score
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palbociclib (Experimental): Palbociclib at a dose of 125 mg once daily, day 1 to day 21 followed by 7 days off treatment in a 28-day cycle for thirteen cycles
  Interventions: Drug: Palbociclib PD-0332991
- Placebo (Placebo Comparator): Placebo of palbociclib once daily day 1 to day 21 followed by 7 days off treatment in a28-day cycle for thirteen cycles
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Palbociclib PD-0332991 — palbociclib at a dose of 125 mg once daily, day 1 to day 21 followed by 7 days off treatment in a 28-day cycle
  Other Names: Ibrance
  Arms: Palbociclib
Drug: Placebo — Arm B: Placebo of palbociclib once daily day 1 to day 21 followed by 7 days off treatment in a 28-day cycle for thirteen cycles
  Arms: Placebo

SUMMARY:
The PENELOPEB study is designed to demonstrate that, in the background of standard anti-hormonal therapy, palbociclib provides superior invasive disease-free survival (iDFS) compared to placebo in pre- and postmenopausal women with HR-positive/HER2-normal early breast cancer at high risk of relapse after showing less than pathological complete response to neoadjuvant taxane- containing chemotherapy. Considering the high risk of recurrence in patients after neoadjuvant chemotherapy and a high CPS-EG score, palbociclib appears to be an attractive option with a favourable safety profile for these patients.

DETAILED DESCRIPTION:
Introduction:

Patients with hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) primary breast cancer who receive chemotherapy as part of their primary treatment are at higher risk of relapse. About a third of the patients with residual invasive disease after neoadjuvant chemotherapy (NACT) will relapse despite adjuvant endocrine therapy (ET). The risk of relapse can be assessed more accurately using the clinical pathological staging-estrogen receptor grading (CPS-EG) scoring system. This involves the tumor stage before treatment start and at surgery, the estrogen receptor (ER) status, and the pathologic grading. A higher score indicates a higher risk of relapse. Patients with a score of three and higher had a disease-free survival of 70% at 5 years despite receiving ET. When combined with the group having a CPS-EG score of two and involved lymph nodes, the disease-free survival increased to 77%. This group comprises about 25% of all patients with residual disease after NACT.

Therapeutic inhibition of cyclin-dependent kinase 4 and 6 (CDK4/6) by palbociclib combined with ET demonstrated clinically relevant efficacy in metastatic HR+ and HER2- breast cancer irrespective of biomarker selection. After the pivotal PALOMA-1 trial, which led to accelerated approval of palbociclib in February 2015, further phase III trials demonstrated that the use of CDK4/6 inhibitors in pre- and postmenopausal patients with hormone-sensitive or resistant cancers, in first-line and pretreated metastatic breast cancer, improves progression-free and overall survival (OS).

Thus, we hypothesized that palbociclib may also be active in patients with residual disease after NACT who are at high risk of relapse. Based on the data from PALOMA-1, we designed the PENELOPE-B trial assessing the efficacy of one year palbociclib vs placebo added to any ET in HR+ and HER2- breast cancer patients with residual disease and high risk after NACT, based on the CPS-EG score.

Patient Selection and Study Design:

PENELOPE-B is a prospective, multicenter, multinational, randomized, double-blind, placebo controlled phase III study investigating the addition of palbociclib for one year to standard adjuvant ET for patients with high-risk residual disease according to the CPS-EG score after NACT for early HR+ and HER2- breast cancer.

The trial was sponsored by GBG Forschungs GmbH in collaboration with NSABP Foundation (plus I-SPY and CCTR), ABCSG, AGO-B, ANBCSG, BIG, Geicam, ICR-CTSU, JBCSG, and KCSG. Pfizer Inc funded the trial and provided drug. The trial was conducted according to ICH-GCP guidelines and the Declaration of Helsinki. The clinical trial Protocol (online only) was approved by the respective health authorities and ethics committees or institutional review boards. All patients provided written informed consent for trial participation, data transfer, and biomaterial collection. The trial was overseen by the International Steering Committee and the GBG Boards and supervised by an Independent Data Monitoring Committee (IDMC).

Eligible patients were randomly assigned in a 1:1 manner in permuted blocks of alternating size 4/6 stratified by risk status (CPS-EG sore ≥ 3 v 2/ypN+), nodal involvement after surgery (ypN0-1 v ypN2-3), Ki-67 (≤ 15% v > 15%), age (≤ 50 v > 50 years), and global region of participating site (Asian v non-Asian).

Treatment:

Patients received either palbociclib 125 mg orally once daily for 21 days followed by 1 week off treatment for a total duration of 13 4-week cycles or matching placebo in addition to standard adjuvant ET at the discretion of the investigator given for at least 5 years. Dose interruptions, reductions, or delays according to predefined toxicity management were acceptable in the case of significant treatment-related toxicity.

Objectives and End Points:

The primary objective of the study was to compare the invasive disease-free survival (iDFS) defined as the time in months between random assignment and first event (ipsilateral invasive in-breast or locoregional recurrence, distant recurrence, invasive contralateral breast cancer, second primary invasive cancer [nonbreast], or death because of any cause) for palbociclib versus placebo. Secondary end points included iDFS excluding second primary invasive nonbreast cancers, distant disease-free survival, OS, locoregional relapse-free interval (LRRFI), safety (which was reported as adverse events (AEs) irrespective of relatedness to study treatment based on National Cancer Institute Common Toxicity Criteria v4.0), and compliance.

All time-to-event end points were analyzed in the intent-to-treat population comprising all randomly assigned patients. Compliance and safety were analyzed in the safety analysis set including all randomly assigned patients who took study medication at least once. For the patients randomly assigned to placebo who received palbociclib at least once during the trial, the treatment group allocation for safety and compliance analyses was the palbociclib arm.

Sample Size and Interim Analyses:

In the initial sample size computation, 233 iDFS events were required to detect a hazard ratio for palbociclib/placebo of 0.67 (from 72% to 80% 3-year iDFS rate) corresponding to a clinically relevant risk reduction of 33% for invasive disease with a power of 85% using a two-sided stratified log-rank test and an overall two-sided significance level of 0.05. Eight hundred patients were planned to be enrolled. To accelerate recruitment after 68 patients had been enrolled, the population was expanded to patients with a CPS-EG score of two and ypN + who were also identified as high-risk patients but with a generally lower risk than the patients with CPS-EG three. Thereafter, the target hazard ratio for palbociclib/placebo was updated to 0.685 (from 77% to 83.6% 3-year iDFS rate), and the iDFS events were increased to 255 and sample size to 1,100 patients.

The study had an adaptive design with two interim efficacy analyses to monitor futility, to test for overwhelming efficacy, and to allow for sample size re-estimation. Safety was assessed at both interim analyses. O'Brien and Fleming type stopping boundaries based on the Lan-DeMets spending function were used in the interim analyses.

Statistical Analysis:

Final analysis of the primary end point iDFS was planned after 290 iDFS events with a nominal significance level of 0.0463 (two-sided). To address the concern of possible inflation of the type I error because of the sample size increase, statistical significance was determined using a weighted statistic of the stratified log-rank test (stratified by risk status, nodal involvement after surgery, Ki-67, age, but not global region of participating site, as prespecified in the Protocol) based on the method of Cui, Hung, and Wang (CHW) with CHW interim monitoring implemented in EAST version 6.5 (Cytel Inc). The 95% repeated CI was reported taking into account the adaptive sample size re-estimation and group sequential nature of the design.

For all other tests, the alpha was set to 0.05 (two-sided). Adjustment for multiple testing in the other tests was not planned. The Kaplan-Meier method was used to estimate the survival probability at specific time points together with a two-sided 95% CI. Univariable Cox-proportional hazards models stratified by the same factors as in the primary analysis were used for time-to-event end points (except LRRFI) to report hazard ratios with 95% CI. LRRFI was analyzed using the cumulative incidence function for rates at specific time points with stratified Gray's test for comparison and stratified univariate Fine-Gray model to report hazard ratio for treatment. Fisher's exact test was used to compare frequencies of AEs between arms.

All statistical analyses were performed using SAS Version 9.4 with SAS Enterprise Guide Version 7.1 on Microsoft Windows 10 Enterprise. Data cutoff date was August 24, 2020.

ELIGIBILITY:
Based on protocol G version 11 dated 09 April 2019

Inclusion Criteria

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Willingness and ability to provide archived formalin fixed paraffin embedded tissue block or a partial block from surgery after neoadjuvant chemotherapy and from core-biopsy before start of neoadjuvant chemotherapy, which will be used for centralized retrospective confirmation of hormone- and HER2-status and to evaluate correlation between genes, proteins, and mRNAs relevant to the endocrine and cell cycle pathways and sensitivity/resistance to the investigational agents. In case of bilateral breast cancer, tumor tissue of both sides needs to be assessable.
3. Histologically confirmed unilateral or bilateral primary invasive carcinoma of the breast.
4. Residual invasive disease post-neoadjuvant either in the breast or as residual nodal invasion.
5. Centrally confirmed hormone-receptor-positive (≥1% ER and/or PR positive stained cells) and HER2-normal (IHC score 0-1 or FISH negative (in-situ hybridization (ISH) ratio) <2.0 status) assessed preferably on tissue from post-neoadjuvant residual invasive disease or core biopsy of the breast, or if no other tissue is available, the residual tumor of the lymph node can be assessed. In case of bilateral breast cancer, hormone receptor positivity and HER2-normal status has to be centrally confirmed for both sides.
6. Centrally assessed Ki-67, pRB, and Cyclin D1 status assessed preferably on post-neoadjuvant residual invasive disease of the breast, or if not possible, of residual nodal invasion or core biopsy. In case of bilateral breast cancer, tumor tissue of both sides needs to be assessable.
7. Patients must have received neoadjuvant chemotherapy of at least 16 weeks. This period must include 6 weeks of a taxane-containing neoadjuvant therapy (Exception: For patients with progressive disease that occurred after at least 6 weeks of taxane-containing neoadjuvant treatment, a total treatment period of less than 16 weeks is also eligible).
8. Adequate surgical treatment including resection of all clinically evident disease and ipsilateral axillary lymph node dissection. Histologically complete resection (R0) of the invasive and ductal in situ tumor is required in case of breast conserving surgery as the final treatment. No evidence of gross residual disease (R2) is required after total mastectomy (R1 resection is acceptable). Axillary dissection is not required in patients with a negative sentinel-node biopsy before (pN0, pN+(mic)) or after (ypN0, ypN+(mic) neoadjuvant chemotherapy.
9. Less than 16 weeks interval since the date of final surgery or less than 10 weeks from completing radiotherapy (whichever occurs last) at date of randomization.
10. Completion of adjuvant radiotherapy according to standard guidelines (e.g. AGO Mamma, NCCN) is strongly recommended. If radiotherapy is not performed, the reason for this needs to be documented in the eCRF.
11. No clinical evidence for locoregional or distant relapse during or after preoperative chemotherapy. Local progression during chemotherapy is not an exclusion criterion.
12. A clinical-pathologic stage - estrogen/grade (CPS-EG) score of ≥3, or score 2 if nodal status at surgery is ypN+, calculated using local estrogen receptor status and grade assessed on either core biopsies taken before start of neoadjuvant treatment or surgical specimen (see chapter 21.1).
13. Age at diagnosis at least 18 years.
14. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
15. Resolution of all acute toxic effects of prior anti cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
16. Estimated life expectancy of at least 5 years irrespective of the diagnosis of breast cancer.
17. The patient must be accessible for scheduled visits, treatment and follow-up. Patients registered in this trial must be treated at the participating center which could be the Principal Investigator's or a Co-investigator's site.

Exclusion Criteria

1. Known severe hypersensitivity reactions to compounds similar to palbociclib or palbociclib/placebo excipients or to endocrine treatments.
2. Inadequate organ function immediate prior to randomization including: Hemoglobin <10g/dL (100g/L); ANC < 2000/mm³ (< 2.0 x 109/L); Platelets <100,000/mm³ (< 100 x 109/L); AST or ALT >1.5 x upper limit of normal (ULN); alkaline phosphatase > 2.5 x ULN, total serum bilirubin > 1.25 x ULN; serum creatinine >1.25 x ULN or estimated creatinine clearance < 60 mL/min as calculated using the method standard for the institution; severe and relevant co-morbidity that would interact with the participation in the study
3. Evidence for infection including wound infections, human immunodeficiency virus (HIV) or any type of hepatitis
4. QTc >480 msec
5. Uncontrolled electrolyte disorders (eg, hypocalcemia, hypokalemia, hypomagnesemia).
6. Any of the following within 6 months of randomization: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 4.0 Grade ≥2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
7. Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or any upper gastrointestinal surgery including gastric resection.
8. Prior malignancy (including invasive or ductal in-situ breast cancer) within 5 years prior to randomization, except curatively treated basal cell carcinoma of the skin and carcinoma in situ of the cervix.
9. Current severe acute or uncontrolled chronic systemic disease (e.g. diabetes mellitus) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
10. Recent (within the past year) or active suicidal behavior.
11. Pregnancy or lactation period. Women of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment and for 90 days after discontinuation. A serum pregnancy test must be negative in premenopausal women or women with amenorrhea of less than 12 months.
12. Major surgery within 2 weeks prior to randomization.
13. 10 weeks or more have passed since completion of radiotherapy at day of randomization and 16 weeks interval since the date of final surgery have passed.
14. Prior treatment with any CDK4/6 inhibitor.
15. Patients treated within the last 7 days prior to randomization and/or concurrent use of drugs known to be strong CYP3A4 inhibitors or inducers
16. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to randomization.
17. Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, MD, Prof, Principal Investigator — ASCO, ESMO, EORTC-TRAFO, ESGO, DKG, AGO
Locations (11):
- NSABP Foundation, Pittsburgh, Pennsylvania, United States
- Contact: Australia and New Zealand Breast Cancer Trials Group, Newcastle, NSW 2310, Australia
- Contact: Austrian Breast & Colorectal Cancer Study Group, Vienna, Austria
- Contact: NSABP Foundation, Multiple Locations, Canada
- Contact: UNICANCER, Paris, France
- Contact: German Breast Group, Neu-Isenburg, Germany
- Contact: Cancer Trials Ireland, Dublin, Ireland
- Contact: Japan Breast Cancer Research Group, Tokyo, Japan
- Contact: Korea Cancer Study Group, Seoul, South Korea
- GEICAM, San Sebastián de los Reyes, Spain
- Contact: Institute of Cancer Research, London, United Kingdom

REFERENCES:
- [Background] Mittendorf EA, Jeruss JS, Tucker SL, Kolli A, Newman LA, Gonzalez-Angulo AM, Buchholz TA, Sahin AA, Cormier JN, Buzdar AU, Hortobagyi GN, Hunt KK. Validation of a novel staging system for disease-specific survival in patients with breast cancer treated with neoadjuvant chemotherapy. J Clin Oncol. 2011 May 20;29(15):1956-62. doi: 10.1200/JCO.2010.31.8469. Epub 2011 Apr 11. PMID 21482989
- [Background] Musgrove EA, Caldon CE, Barraclough J, Stone A, Sutherland RL. Cyclin D as a therapeutic target in cancer. Nat Rev Cancer. 2011 Jul 7;11(8):558-72. doi: 10.1038/nrc3090. PMID 21734724
- [Background] ENCODE Project Consortium. An integrated encyclopedia of DNA elements in the human genome. Nature. 2012 Sep 6;489(7414):57-74. doi: 10.1038/nature11247. PMID 22955616
- [Background] Finn RS, Dering J, Conklin D, Kalous O, Cohen DJ, Desai AJ, Ginther C, Atefi M, Chen I, Fowst C, Los G, Slamon DJ. PD 0332991, a selective cyclin D kinase 4/6 inhibitor, preferentially inhibits proliferation of luminal estrogen receptor-positive human breast cancer cell lines in vitro. Breast Cancer Res. 2009;11(5):R77. doi: 10.1186/bcr2419. PMID 19874578
- [Background] Symmans WF, Peintinger F, Hatzis C, Rajan R, Kuerer H, Valero V, Assad L, Poniecka A, Hennessy B, Green M, Buzdar AU, Singletary SE, Hortobagyi GN, Pusztai L. Measurement of residual breast cancer burden to predict survival after neoadjuvant chemotherapy. J Clin Oncol. 2007 Oct 1;25(28):4414-22. doi: 10.1200/JCO.2007.10.6823. Epub 2007 Sep 4. PMID 17785706
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Result] Loibl S, Marme F, Martin M, Untch M, Bonnefoi H, Kim SB, Bear H, McCarthy N, Mele Olive M, Gelmon K, Garcia-Saenz J, Kelly CM, Reimer T, Toi M, Rugo HS, Denkert C, Gnant M, Makris A, Koehler M, Huang-Bartelett C, Lechuga Frean MJ, Colleoni M, Werutsky G, Seiler S, Burchardi N, Nekljudova V, von Minckwitz G. Palbociclib for Residual High-Risk Invasive HR-Positive and HER2-Negative Early Breast Cancer-The Penelope-B Trial. J Clin Oncol. 2021 May 10;39(14):1518-1530. doi: 10.1200/JCO.20.03639. Epub 2021 Apr 1. PMID 33793299
- [Derived] Hahnen E, Hauke J, Gelmon K, Marme F, Ernst C, Martin M, Untch M, Bonnefoi H, Knudsen E, Im SA, DeMichele A, Van't Veer L, Kim SB, Bear H, McCarthy N, Rhiem K, Turner N, Witkiewicz A, Rojo F, Filipits M, Martin LA, Fasching PA, Schem C, Becker K, Garcia-Saenz JA, Kelly CM, Reimer T, Toi M, Rugo HS, Denkert C, Gnant M, Makris A, Liu Y, Valota O, Felder B, Weber K, Nekljudova V, Loibl S. BRCA1/2 and Other Predisposition Genes in High-Risk Hormone Receptor+/Human Epidermal Growth Factor Receptor 2- Breast Cancer Treated With Endocrine Therapy With or Without Palbociclib: A Secondary PENELOPE-B Study Analysis. JCO Precis Oncol. 2025 Apr;9:e2400742. doi: 10.1200/PO-24-00742. Epub 2025 Apr 10. PMID 40209141
- See also: General trial information — http://www.gbg.de/en/trials/penelope.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 4 years (Q-I 2014 -Q-IV 2017) in 221 sites worldwide (11 countries). 1708 patients were screened, 1250 patients were randomized (Palbociclib 631; Placebo 619).
Pre-assignment Details: Female patients >=18 years with residual invasive disease after NACT (in breast or lymph nodes), centrally assessed ER+ and/or PgR+ and HER2- tumors and centrally assessed Ki-67 status and a CPS-EG score of >=3 or 2 with ypN1 (after amendment 3, February 9, 2015) were eligible. >=16weeks NACT (incl. 6 weeks taxane), surgery and radiation received.
Period: Overall Study
Arm/Group | Palbociclib | Placebo
Started (Randomly assigned to each arm) | 631 | 619
Started Treatment (Started treatment in each arm) | 628 | 616
Safety Population (N=5 patients who started treatment with placebo received palbociclib once; hence, they were analyzed for safety in the palbociclib arm.) | 633 | 611
Completed | 508 | 523
Not Completed | 123 | 96
Not completed — Disease recurrence | 25 | 40
Not completed — Second primary invasive nonbreast | 2 | 3
Not completed — Death | 2 | 1
Not completed — Adverse Event | 33 | 5
Not completed — Withdrawal by Subject | 56 | 41
Not completed — Physician Decision | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib | Placebo | Total
Number analyzed (Participants) | 631 | 619 | 1250
Age, Continuous [Median (Full Range); unit: years] | 49 [22 to 76] | 48 [19 to 79] | 49 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 631 | 619 | 1250
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG performance status [Count of Participants; unit: Participants] — ECOG 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG 0 | 537 | 527 | 1064
    ECOG 1 | 94 | 92 | 186
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 300 | 316 | 616
  Postmenopausal | 331 | 303 | 634

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease Free Survival (iDFS) for Palbociclib vs. Placebo in Patients With High CPS-EG Score After Neoadjuvant Chemotherapy Receiving Standard Adjuvant Endocrine Therapy for HR-positive/HER2-normal Primary Breast Cancer.
Description: Invasive disease-free survival (iDFS) is defined according to Hudis (J Clin Oncol 2007) as the time period between randomization and first event (ipsi- or contralateral invasive in-breast or loco-regional recurrence, distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause, invasive contralateral breast cancer, second primary invasive cancer (non-breast)) assessed until the end of study.
Time Frame: From date of randomisation to data cut off: 24 August 2020 (approximately 6 years and 6 months)
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: % of patients without invasive disease
Arm/Group | Palbociclib | Placebo
Number analyzed (Participants) | 631 | 619
% of patients without invasive disease
  3-year iDFS | 81.2 [77.8 to 84.1] | 77.7 [74.1 to 80.9]
  5-year iDFS | 63.6 [56.4 to 69.9] | 67.9 [61.6 to 73.3]

2. Secondary Outcome: iDFS Excluding Second Non-breast Cancers
Description: Invasive disease-free survival (iDFS) is defined according to Hudis (J Clin Oncol 2007) as the time period between randomization and first event assessed until the end of study.
Time Frame: From date of randomisation to data cut off: 24 August 2020 (approximately 6 years and 6 months)
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: % of patients free of event
Arm/Group | Palbociclib | Placebo
Number analyzed (Participants) | 631 | 619
% of patients free of event
  3-year iDFS | 82 [78.6 to 84.9] | 78.5 [75 to 81.7]
  5-year iDFS | 64 [56.6 to 70.4] | 68.6 [62.4 to 74.1]

3. Secondary Outcome: Distant Disease Free Survival (DDFS)
Description: Distant disease free survival (DDFS) is defined as the time period between randomization and diagnosis of first distant breast cancer recurrences assessed until the end of study.
Time Frame: From date of randomisation to data cut off: 24 August 2020 (approximately 6 years and 6 months)
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: % of patients free of event
Arm/Group | Palbociclib | Placebo
Number analyzed (Participants) | 631 | 619
% of patients free of event
  3-year DDFS | 82.4 [79.1 to 85.3] | 80 [76.6 to 83.1]
  5-year DDFS | 65.8 [58.5 to 72.1] | 69.9 [63.8 to 75.2]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time period between randomization and death of any cause assessed until the end of study.
Time Frame: From date of randomisation to data cut off: 24 August 2020 (approximately 6 years and 6 months)
Population: Intention-to-treat analysis
Measure: Number (95% Confidence Interval); unit: % of patients free of event
Arm/Group | Palbociclib | Placebo
Number analyzed (Participants) | 631 | 619
% of patients free of event
  3-year OS | 93.6 [91.3 to 95.3] | 90.5 [87.8 to 92.6]
  5-year OS | 79.6 [72.1 to 85.3] | 84.6 [78.9 to 88.9]

ADVERSE EVENTS:
Time Frame: For AEs and SAEs, the reporting period is from the time the patient took the first dose of the investigational product until (and including) 30 calendar days after the last administration of the investigational product (i.e., from first dose to 30 days after last dose). Serious and Other (Not Including Serious) Adverse Events were assessed for up to 14 months, and all-cause mortality was assessed up to 6 years and 6 months.
Description: All recorded events meeting the definitions of All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events are currently reported.
Arm/Group | Palbociclib | Placebo
All-Cause Mortality (participants affected / at risk) | 63/633 | 67/611
Serious Adverse Events (participants affected / at risk) | 64/633 | 65/611
Other Adverse Events (participants affected / at risk) | 632/633 | 610/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib (N=633) | Placebo (N=611)
Infections and infestations (Infections and infestations) | 19 | 25
Cellulitis (Infections and infestations) | 4 | 5
Erysipelas (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 3 | 1
Postoperative wound infection (Infections and infestations) | 0 | 3
Wound infection (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 | 10
Overdose (Injury, poisoning and procedural complications) | 7 | 3
Fracture (Injury, poisoning and procedural complications) | 2 | 2
Seroma (Injury, poisoning and procedural complications) | 2 | 0
Vascular disorders (Vascular disorders) | 6 | 4
Pulmonary embolism (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 0 | 2
General disorders and administration site conditions (General disorders) | 3 | 4
Impaired healing (General disorders) | 1 | 1
Nervous system disorders (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 1 | 1
Blood and the lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Musculoskeletal, connective tissue and bone disorders (Musculoskeletal and connective tissue disorders) | 3 | 2
Neoplasms benign and malignant (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Gastrointestinal disorders (Gastrointestinal disorders) | 3 | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hepato-biliary disorders (Hepatobiliary disorders) | 0 | 3
Psychiatric disorders (Psychiatric disorders) | 1 | 2
Renal and urinary disorders (Renal and urinary disorders) | 3 | 0
Cardiac disorders (Cardiac disorders) | 2 | 0
Eye disorders (Eye disorders) | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
Surgical and medical procedures (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib (N=633) | Placebo (N=611)
Hot flush (Vascular disorders) | 277 | 311
Hypertension (Vascular disorders) | 54 | 60
Embolism (Vascular disorders) | 13 | 7
Fatigue (General disorders) | 420 | 312
Peripheral edema (General disorders) | 126 | 99
Pyrexia (General disorders) | 71 | 49
Vaginal dryness (Reproductive system and breast disorders) | 52 | 55
Vaginal hemorrhage (Reproductive system and breast disorders) | 12 | 15
Alanine aminotransferase increased (Investigations) | 138 | 141
Aspartate aminotransferase increased (Investigations) | 131 | 102
Blood alkaline phosphatase increased (Investigations) | 106 | 120
Blood creatinine increased (Investigations) | 78 | 67
Blood albumin decreased (Investigations) | 63 | 46
Blood bilirubin increased (Investigations) | 42 | 44
Leukopenia (Blood and lymphatic system disorders) | 628 | 427
Neutropenia (Blood and lymphatic system disorders) | 606 | 143
Anemia (Blood and lymphatic system disorders) | 468 | 185
Thrombocytopenia (Blood and lymphatic system disorders) | 358 | 99
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 132 | 99
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 73 | 43
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 | 8
Dysgeusia (Nervous system disorders) | 41 | 32
Headache (Nervous system disorders) | 147 | 141
Other nervous system disorders (Nervous system disorders) | 133 | 138
Cataract (Eye disorders) | 6 | 7
Vertigo (Ear and labyrinth disorders) | 46 | 43
Nausea (Gastrointestinal disorders) | 150 | 126
Stomatitis (Gastrointestinal disorders) | 174 | 53
Constipation (Gastrointestinal disorders) | 140 | 84
Diarrhea (Gastrointestinal disorders) | 116 | 96
Vomiting (Gastrointestinal disorders) | 66 | 57
Abdominal distension (Gastrointestinal disorders) | 17 | 21
Other gastrointestinal disorders (Gastrointestinal disorders) | 147 | 107
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 175 | 145
Arthralgia (Musculoskeletal and connective tissue disorders) | 261 | 286
Myalgia (Musculoskeletal and connective tissue disorders) | 128 | 113
Bone pain (Musculoskeletal and connective tissue disorders) | 109 | 117
Other nusculoskeletal, connective tissue and bone disorders (Musculoskeletal and connective tissue disorders) | 122 | 133
Hypocalcemia (Metabolism and nutrition disorders) | 223 | 149
Hypomagnesemia (Metabolism and nutrition disorders) | 186 | 173
Hyperkalemia (Metabolism and nutrition disorders) | 67 | 80
Hypernatremia (Metabolism and nutrition disorders) | 57 | 52
Hyponatremia (Metabolism and nutrition disorders) | 47 | 41
Hypokalemia (Metabolism and nutrition disorders) | 52 | 30
Decreased appetite (Metabolism and nutrition disorders) | 51 | 29
Hypercalcemia (Metabolism and nutrition disorders) | 20 | 27
Glucose tolerance impaired (Metabolism and nutrition disorders) | 14 | 14
Infection (Infections and infestations) | 379 | 312

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Only after the sponsor's publication of the overall study results of the primary endpoint do participating sites have the right to publish publications related to study data collected by participating sites, and any results of add-on research conducted by participating sites, subject to compliance with the study publications and presentations policy.

DOCUMENTS (3):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT01864746/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT01864746/SAP_001.pdf
  • Informed Consent Form (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT01864746/ICF_002.pdf